CLINICAL TRIAL: NCT06318936
Title: RSV Burden in Older Adults in Primary Care in The Netherlands: the RAPID Study
Brief Title: Respiratory Syncytial Virus (RSV) Burden in Older Adults in Primary Care in The Netherlands
Acronym: RAPID
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Janssen-Cilag B.V. (Industry)
Responsible Party: Principal Investigator, Louis Bont, Prof. dr. Louis Bont, UMC Utrecht
Other Study IDs: 22-677
Record Dates: First submitted 2024-01-21; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: RSV Infection
Keywords: older adults; RSV; burden; outpatient; primary care
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults with RSV infection: Adults aged ≥60 years attending primary care with acute respiratory tract infecion

SUMMARY:
RSV infection is a leading cause of medical care in older adults, sometimes leading to hospital admission and severe outcomes. Although the majority of RSV infections are managed outside hospitals, little is known on the burden of RSV in older adults in the primary care setting. Accurate estimates of the RSV burden in primary care is particularly relevant since vaccines against RSV infection in older adults will likely become available for the general population soon. The use of high-quality point-of-care (POC) molecular viral diagnostics allows to identify RSV infected older adults and would therefore contribute to fill one of the most important gaps in knowledge facilitating implementation of RSV vaccination of older adults

With this prospective, observational study, we aim to define the disease burden of RSV infection in older adults in the primary care setting.

DETAILED DESCRIPTION:
Th RAPID study is a prospective, observational study in Dutch primary care practices during two RSV seasons. As part of routine care, rapid molecular viral diagnostic testing on respiratory samples will be offered to all older adults attending the primary care physician because of symptoms of acute respiratory tract infection (ARTI). RSV positive cases will be included for further study. Participants will be asked to fill out three questionnaires by phone or by online at day 0, 14 and 30 after the GP-visit.

The main endpoint is the burden of medically attended RSV infection in the Dutch primary care setting, quantified using several clinical and socioeconomic parameters, including (but not limited to) clinical symptoms and their duration, medicine use, hospitalisation rate, quality of life and ability to perform normal daily activities. Secondary, data on health care consumption and indirect costs will be collected and we will assess the effect of age and severe comorbidity on clinical course of RSV disease.

A population size of 1000 older adults age >60 years presenting with acute respiratory symptoms to the general practitioner (GP) during RSV season will be tested for RSV as part of routine care. We expect about 100 RSV+. Based on our sample size calculation, 100 RSV+ cases would provide sufficient accuracy for estimating the relevant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age (≥60 years of age)
* RSV positive
* Subject is willing and able to give informed consent for participation in the study
* Subject is willing and able to adhere to protocol-specific procedures

Exclusion Criteria:

* Subject is not able to understand and communicate in the local language or English.
* Previous or current participation in RSV interventional trial (vaccine, antivirals)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All older adults (≥60 years of age) who visit their general practitioner because of acute respiratory tract symptoms such as shortness of breath, cough, sore throat or coryza (WHO definition) in one of the participating primary care practices in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Burden of medically attended RSV infection in the Dutch primary care | Data will be collected at three timepoints (Day 0, Day 14 and Day 30 days after viral swab)
  The burden of medically attended RSV infection in the Dutch primary care setting will be defined as severity and duration of clinical symptoms, and healthcare resource use.

SECONDARY OUTCOMES:
RSV-related health care consumption and indirect costs in older adults | Data will be collected at three timepoints (Day 0, Day 14 and Day 30 days after viral swab)
  Health care utilization will be calculated as the number of contact moments (including phone contacts, telemedicine and visits) with the GP-practices and other health-care providers (e.g. visit to specialist, emergency department). For hospitalized adults, the number of admitted days and the level of care (general ward, high dependency unit, intensive care unit) will be calculated.
  Medical costs and socio-economic costs will be calculated based on the questionnaires at day 0, 14 and day 30.
Proportion of medically attended RSV infection amongst all medically attended acute respiratory infections in older adults in the primary care setting | At day of sampling (Day 0)
  The proportion of RSV positive older adults will be calculated as the number of older adults who tested positive for RSV divided by the total number of older adults who visit the participating GP practices because of ARTIs and were tested for RSV.
Association between disease severity and several clinical and demographic parameters (e.g. age, cardiopulmonary comorbidity, smoking status, chronic immunosuppressive medication use) and RSV burden (by disease severity and healthcare usage) | Data will be collected at three timepoints (Day 0, Day 14 and Day 30 after viral swab)
  We will explore potential risk factors ((e.g. age, cardiopulmonary comorbidity, smoking status, polypharmacy, chronic immunosuppressive medication use) for severe RSV disease.
Incidence of RSV-related secondary bacterial pneumonia events and antibiotic use | Data will be collected at the last timepoint (30 days after viral swab)
  Incidence will be calculated as the proportion of subjects that show RSV-associated secondary bacterial pneumonia events (defined as pneumonia within 21 days after RSV infection) and antibiotic use.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bont, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands